CLINICAL TRIAL: NCT01044784
Title: Acute Evaluation of the Safety of LV-LV Delays and Its Effects on Mechanical Dyssynchrony
Brief Title: Acute Evaluation of the Safety of Left Ventricular-left Ventricular (LV-LV) Delays and Its Effects on Mechanical Dyssynchrony
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 60028011
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Resynchronization Therapy
Keywords: CRT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the effects of various LV-LV delays during multi-site left ventricular (MSLV) pacing on mechanical dyssynchrony in cardiac resynchronization therapy (CRT) patients post-implant.

ELIGIBILITY:
Inclusion Criteria:

1. Have an approved indication for a CRT implant
2. Undergoing or previously received the implant of a St. Jude Medical Promote Q 3221-36 CRT-D with a Quartet Model 1458Q LV lead at participating clinical study site
3. Ability to provide informed consent for study participation and be willing and able to comply with the prescribed evaluations

Exclusion Criteria:

1. Have persistent or permanent atrial fibrillation
2. Have an intrinsic heart rate of <50 beats per minute
3. Have Cheyne-Stokes breathing
4. Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures
5. Have had a recent CVA or TIA within 3 months prior to enrollment
6. Be less than 18 years of age
7. Be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for standard CRT-D indications.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Schuchtermannklinik, Bad Rothenfelde, Germany

REFERENCES:
- [Derived] Rinaldi CA, Leclercq C, Kranig W, Kacet S, Betts T, Bordachar P, Gutleben KJ, Shetty A, Donal E, Keel A, Ryu K, Farazi TG, Simon M, Naqvi TZ. Improvement in acute contractility and hemodynamics with multipoint pacing via a left ventricular quadripolar pacing lead. J Interv Card Electrophysiol. 2014 Jun;40(1):75-80. doi: 10.1007/s10840-014-9891-1. Epub 2014 Mar 14. PMID 24626999
- [Derived] Rinaldi CA, Kranig W, Leclercq C, Kacet S, Betts T, Bordachar P, Gutleben KJ, Shetty A, Keel A, Ryu K, Farazi TG, Simon M, Naqvi TZ. Acute effects of multisite left ventricular pacing on mechanical dyssynchrony in patients receiving cardiac resynchronization therapy. J Card Fail. 2013 Nov;19(11):731-8. doi: 10.1016/j.cardfail.2013.10.003. Epub 2013 Oct 10. PMID 24263116